CLINICAL TRIAL: NCT00756327
Title: AquaLase Capsule Wash for Pediatric Eyes
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Rupalben Trivedi, MD, Medical University of South Carolina
Other Study IDs: MRC-08-001
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Cataract; Pediatric Cataract
Keywords: pediatric eyes; bilateral cataract; IOL implantation; Aqualase capsule wash; posterior capsule opacification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
To determine whether AquaLase capsule wash reduces posterior capsule opacification (PCO) in pediatric eyes.

DETAILED DESCRIPTION:
Dramatic advances have occurred in the treatment of childhood cataracts in the last 10 years. Intraocular lens (IOL) implantation has been universally accepted as the standard of care for most children undergoing cataract surgery beyond infancy. Despite advances in cataract surgery in children, PCO remained a significant complication following pediatric cataract surgery. In addition to being visually disturbing, it also induces amblyopia in children and if not treated at the earliest, irreversible visual changes may occur. The younger the child, the more acute is the problem: PCO occurs faster and the effect of amblyopia is more pronounced.

To prevent opacification of the visual axis after cataract surgery, primary posterior capsulectomy and vitrectomy are routinely needed while managing pediatric cataract. This surgical step is not routinely used in adult cataract surgery, where we prefer an intact posterior capsule. Researchers are constantly trying to find a way to avoid the need for invasive procedures like posterior capsulectomy and vitrectomy for pediatric eyes. Use of AquaLase technology has shown some capability in cleaning the capsular bag during cataract surgery. Observations of this include anecdotal observation from users. AquaLase for cataract removal with the Infiniti Vision System has been used since 2003, is registered, and the FDA clearance is 510(k) number K980292. AquaLase uses pulses of warmed balanced salt solution to gently emulsify and facilitate aspiration of cataracts. The device under evaluation falls under the same FDA clearance. The unique aspect is the application tip which is intended to allow more thorough capsular bag cleaning or removal of more residual lens material than is currently being achieved. The energy source, controls, and materials are all identical to the currently marketed product. The difference is in the geometry of the distal most end of the application tip.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataract in a child aged 6-15 years old
* Informed consent from the parents/legal guardian.

Exclusion Criteria:

* traumatic cataract
* fellow eye - visually not significant cataract
* fellow eye surgery not scheduled within 3-month period after first eye surgery
* dense posterior capsule plaque
* preexisting posterior capsule defect
* subluxated cataract
* high myopia (defined as axial length >24 mm)
* child with multiple disability where it may not be feasible to perform YAG laser capsulotomy in the office, if needed
* Participants with a strong likelihood of non-adherence (difficulties in adhering to follow-up schedule due to geographic distance from clinical center)

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with bilateral cataract undergoing surgery for cataract aspiration and IOL implantation. Bilateral cataract in a child aged 6-15 years old.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trivedi Rupalben, MD, Principal Investigator — Assistant Professor
Locations (1):
- Aravind Haripriya, Madurai, India